CLINICAL TRIAL: NCT03594487
Title: Fecal Microbiota Transplantation (FMT) of FMP30 in Relapsing-Remitting Multiple Sclerosis: A Phase 1b Clinical Trial to Evaluate Feasibility, Safety, Tolerability and Effects on Immune Function
Brief Title: Fecal Microbiota Transplantation (FMT) of FMP30 in Relapsing-Remitting Multiple Sclerosis
Acronym: MS-BIOME
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Under-enrollment, including after interruption due to a hold on source FMT material and the COVID-19 pandemic
Sponsor: Jeffrey Gelfand (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Gelfand, Professor of Clinical Neurology, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-23827
Record Dates: First submitted 2018-06-07; First posted 2018-07-20 (Actual); Results first posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Relapsing Remitting Multiple Sclerosis; Fecal Microbiota Transplantation
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Interventional FMT Treatment Arm (Experimental): After providing written informed consent, participants will undergo screening and baseline assessments of stool and blood sampling, questionnaires, physical examination, MS rating scales, and MRI. Participants will then initiate an oral antibiotic regimen for 5 days to precondition the gut for the Fecal Microbiota Transplantation (FMT) of FMP30 donor stool and optimize engraftment of the FMP30 donor stool microbiome. Following standard bowel preparation for colonoscopy, participants will undergo the FMT procedure by an experienced gastroenterologist. Participants will return for scheduled assessments and follow-up MRI for 12 weeks, with additional safety and biomarker follow-up for 36 weeks.
  The active study time is designed to be short (12 weeks active phase) to minimize time off on other MS disease-modifying therapy (DMT). This arm of the study will last for approximately 52 weeks total (4 weeks of screening + 12 weeks active treatment phase + 36 weeks of safety follow-up).
  Interventions: Drug: FMP30 Donor Stool; Procedure: Fecal Microbiota Transplantation (FMT) of FMP30 Donor Stool
- Observational Control Arm (Active Comparator): Participants, who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration, and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures.
  After providing written informed consent, participants will undergo screening and baseline assessments, including collection of blood and stool samples, demographic data collection, concomitant medication review, and an MS Relapse assessment. At week 2, participants will mail in stool samples with a prepaid air bill and packaging. Weeks 4, 8, and 12 assessments will include concomitant medication review, relapse assessment, and blood and stool collection.
  The duration of the study for the observational control arm will last for 12 weeks. All study procedures will be performed at the University of California, San Francisco.
  Interventions: Other: Observational Control

INTERVENTIONS:
Drug: FMP30 Donor Stool — FMP30 is manufactured by the non-profit stool bank Openbiome. Each FMP30 filtered donor stool engraftment has approximately 12.5g of stool per 30mL of normal saline. It is homogenized in sterile normal saline.
  Arms: Interventional FMT Treatment Arm
Procedure: Fecal Microbiota Transplantation (FMT) of FMP30 Donor Stool — Three doses of filtered donor stool engraftments homogenized in sterile normal saline (FMP30), obtained from the non-profit stool bank OpenBiome, will be administered via colonoscopy in patients with Relapsing-Remitting Multiple Sclerosis. FMT dosage via colonoscopy may include a lower amount of transplanted stool at the discretion of the study gastroenterologist if there are any peri-procedural safety or technical considerations. Total FMT dose (in milliliters) will be documented.
  Arms: Interventional FMT Treatment Arm
Other: Observational Control — Participants, who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration, and prior use of allowable MS therapies will be recruited as a comparison observational group to measure stability of stool and serum immunological measures.
  Arms: Observational Control Arm

SUMMARY:
In this Phase 1b open-label prospective clinical trial, patients with relapsing-remitting MS will undergo FMT of FMP30 (donor stool) via colonoscopy and immunological efficacy endpoints will be assessed at various time points. The active phase of the study will continue for 12 weeks post-FMT with safety and biomarker (engraftment) follow-up for 48 weeks. A parallel observational control arm of MS patients who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures. The study duration for the Observational Control Arm is 12 weeks.

DETAILED DESCRIPTION:
In this Phase 1b open-label prospective clinical trial, patients with relapsing- remitting MS will undergo FMT of FMP30 (donor stool) via colonoscopy and immunological efficacy endpoints will be assessed at various time points. The active phase of the study will continue for 12 weeks post-FMT with safety and biomarker (engraftment) follow-up for 48 weeks. A parallel observational control arm of MS patients who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures.

The primary hypotheses are that:

1. FMT will be safe and tolerable in patients with MS.
2. FMT preceded by antibiotic preconditioning will lead to a change in fecal microbiota community structure.

Secondary hypotheses are that:

1. FMT preceded by antibiotic preconditioning will induce a favorable shift from pro-inflammatory to immunomodulatory T cell profiles in patients with relapsing-remitting MS.
2. That engraftment will not appreciably decay over time.
3. That FMT will favorably change humoral function.
4. That FMT will favorably influence short-term clinical and radiological endpoints.

FMP30 donor stool will be obtained from OpenBiome (Somerville, Massachusetts; OpenBiome.org), an established nonprofit stool bank with stringent safety protocols and quality control. Donor stool will be obtained from donors without Multiple Sclerosis (MS) and without other known autoimmune diseases and will be screened for transmissible pathogens. In collaboration with OpenBiome, University of California, San Francisco (UCSF) will additionally screen donor stool using in vitro assays for immunological properties thought to be favorable in Multiple Sclerosis (MS), including decreasing T helper 17 cells (TH17) and increasing T regulatory cells, in order to select the final donor stool to be used in this study for FMT. UCSF will obtain an investigational new drug (IND) from the FDA for FMT of FMP30 donor stool in MS.

After providing written informed consent and reviewing inclusion and exclusion criteria, participants will participate in either the FMT Treatment Arm or the Observational Control Arm.

Participants in the FMT Treatment Arm will first undergo screening assessments according to the study schedule of activities and provide blood samples for eligibility and research, and stool samples for research. Participants who pass screening will have their pre-treatment baseline visit with 21 days of their screening visit where they will have an MRI, safety and biomarker research blood sample collection, stool sample collection for research, complete study activities according to the study visit schedule, be given antibiotics, bowel preparation, a medication compliance diary and directions on when and how to start the antibiotics and bowel preparation before their scheduled FMT colonoscopy procedure.

The week before their Baseline FMT visit, participants will be contacted by study staff to initiate an oral antibiotic regimen for 5 days to precondition the gut for FMT and optimize engraftment of the donor microbiome. Study staff will ensure that the participants understand how to complete their oral antibiotic regimen, compliance diary, and bowel preparation correctly.

At the study Baseline Visit, following standard bowel preparation for colonoscopy, participants will then undergo colonoscopy with FMT of FMP30 by an experienced gastroenterologist. Participants will return for scheduled assessments of stool and blood sampling, questionnaires, physical examination, MS rating scales, and follow-up MRI for 12 weeks, with additional safety and biomarker blood sample collection, and followed at weeks 24, 36, and 48. The active study time of 12 weeks was designed to be short to minimize time off MS disease-modifying therapies (should the participant wish to go on a MS disease-modifying therapy).

Participants participating in the Observational Control Arm will not undergo the interventional FMT treatment. Participants in this arm will have a total of 5 visits over the course of 12 weeks. At the Screening/Baseline visit, participants will provide blood and stool samples for research along with other study activities, according to the study visit schedule. Participants will mail in a stool sample at week 2 and come in for follow-up visits at weeks 4, 8, and 12.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 inclusive (at time of screening).
2. Diagnosis of relapsing-remitting multiple sclerosis (MS) by the International Panel McDonald Criteria (2010)(1), incorporating 2017 revisions, which reclassify select high-risk Clinically Isolated Syndromes under 2010 criteria as RRMS under 2017 criteria, and Lublin criteria (2014)(2). [RRMS: relapsing remitting multiple sclerosis]
3. Recent documented MS disease activity, defined as at least 1 clinical relapse within the past 1 year prior to baseline OR 2 clinical relapses in the past 2 years prior to baseline OR at least 1 new T2/FLAIR lesion on brain or spine MRI OR at least 1 gadolinium enhancing lesion on brain or spine MRI in the past 1 year prior to baseline.
4. Expanded Disability Status Scale (EDSS) less than or equal to 6.0; EDSS 5.5 or less if MS disease duration is greater than 15 years (no other disease duration restriction).
5. Must have positive serology for Epstein-Barr Virus (EBV) (IgG anti-EBNA positive) at screening, indicating prior exposure. [EBNA: Epstein-Barr nuclear antigen]
6. No prior MS disease-modifying therapy or a 12-week washout period for participants on glatiramer acetate or interferon-beta therapy.
7. At least 4 weeks from baseline since last use of IV or oral glucocorticoids. Protocol: MS-BIOME Study.
8. Agree to maintain a stable diet during the course of the study (over-the-counter probiotics are allowable).
9. Premenopausal women and women <12 months after the onset of menopause must have a negative serum pregnancy test unless they have undergone surgical sterilization.
10. Female participants of childbearing potential who are sexually active with a non-sterilized male partner must agree to use a highly effective method of contraception; non-sterilized male participants who are sexually active with a female partner of childbearing potential must agree to use a highly effective method of contraception.
11. Not actively participating in another interventional MS clinical trial (participation in other observational research studies is allowable).

Exclusion Criteria:

1. Prior use of fingolimod, dimethyl fumarate, teriflunomide, natalizumab, alemtuzumab, mitoxantrone, cyclophosphamide, rituximab, ocrelizumab, daclizumab, methotrexate, azathioprine, mycophenolate mofetil, cyclosporine, leflunomide, or induction chemotherapy.
2. No use of diuretics like furosemide (Lasix) 1 week before the first dose of oral antibiotics. The use of hydrochlorothiazide (HCTZ) for hypertension at a dose < 50 mg/day is allowable.
3. Progressive MS by Lublin criteria (2014).
4. No oral or IV antibiotics are allowed within 8 weeks prior to screening and within 12 weeks prior to the planned FMT procedure (for participants in the FMT arm) or prior to the first stool collection (for participants in the control arm). (Note that topical, otic, ocular antibiotics are specifically allowable, which is consistent with the IMSMS.org protocol for collaborative gut microbiome research in MS). [IMSMS: International MS Microbiome Study]
5. Hypersensitivity or allergy to study antibiotics, conscious sedation medications, or bowel preparation.
6. Contraindication to study procedures, including MRI, anesthesia (ASA criteria IV and V), colonoscopy, and phlebotomy.
7. History of inflammatory bowel disease (Crohn's Disease, Ulcerative Colitis) Protocol: MS-BIOME Study.
8. Active symptomatic C. Difficile infection (colonization is not an exclusion).
9. Active gastrointestinal condition being investigated (i.e. GI bleeding, colon cancer, active GI workup); history of known or suspected toxic megacolon and/or known small bowel ileus, major gastrointestinal surgery (e.g. significant bowel resection) within 3 months before enrollment (note that this does not include appendectomy or cholecystectomy); or history of total colectomy or bariatric surgery.
10. History of malignancy (except excised cutaneous basal cell carcinoma or squamous cell carcinoma, which are allowable), including no concurrent induction chemotherapy, radiation therapy, or biological treatment for active malignancy.
11. Pregnant or lactating women or intention of getting pregnant during the trial period.
12. Active infection, including untreated latent or active tuberculosis, HIV, hepatitis, syphilis, or other major active infection.
13. Known immunodeficiency, including Common Variable Immunodeficiency (CVID).
14. INR>1.5, Platelets<100, Hemoglobin <8.5, WBC<2.0, Absolute lymphocyte count <0.8, Absolute Neutrophil Count <0.5, CD4<200, eGFR<45. [INR: international normalized ratio, WBC: White Blood cell, CD4: cluster of differentiation 4, eGFR: epidermal growth factor receptor]
15. Any condition that in the opinion of the study PI could jeopardize the safety of the participant, would make it unlikely for the participant to complete the study or could confound the results of the study.
16. Unable or unwilling to comply with study protocol requirements.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Gelfand, MD, MAS, Principal Investigator — UCSF Multiple Sclerosis Center
Locations (1):
- UCSF Multiple Sclerosis Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Outcome data as well as study data related to diagnosis, disease presentation, and date of birth, along with biological specimens collected as part of the study, may be shared (in coded form) in the future with other qualified researchers on a case by case basis at the discretion of the PI and Co-PIs. Any such investigator will be required to provide appropriate documentation that the research being conducted has been approved by an Institutional Review Board and demonstrate that it will be of value in determining the cause of MS or a related disorder, and as allowed by the UCSF Institutional Review Board.
Supporting Information: Study Protocol
Time Frame: After initial study results are published and on a case by case basis.
Access Criteria: Limited data to include demographic and clinical information and biological specimens collected as part of the study, may be shared (in coded form) in the future with other qualified researchers on a case by case basis at the discretion of the PI and Co-PIs. Any such investigator will be required to provide appropriate documentation that the research being conducted has been approved by an Institutional Review Board and demonstrate that it will be of value in determining the cause of MS or a related disorder, and as allowed by the UCSF Institutional Review Board.

REFERENCES:
- [Background] Cekanaviciute E, Yoo BB, Runia TF, Debelius JW, Singh S, Nelson CA, Kanner R, Bencosme Y, Lee YK, Hauser SL, Crabtree-Hartman E, Sand IK, Gacias M, Zhu Y, Casaccia P, Cree BAC, Knight R, Mazmanian SK, Baranzini SE. Gut bacteria from multiple sclerosis patients modulate human T cells and exacerbate symptoms in mouse models. Proc Natl Acad Sci U S A. 2017 Oct 3;114(40):10713-10718. doi: 10.1073/pnas.1711235114. Epub 2017 Sep 11. PMID 28893978
- [Background] Bafeta A, Yavchitz A, Riveros C, Batista R, Ravaud P. Methods and Reporting Studies Assessing Fecal Microbiota Transplantation: A Systematic Review. Ann Intern Med. 2017 Jul 4;167(1):34-39. doi: 10.7326/M16-2810. Epub 2017 May 23. PMID 28531908
- [Background] Morris MS, Graham LA, Chu DI, Cannon JA, Hawn MT. Oral Antibiotic Bowel Preparation Significantly Reduces Surgical Site Infection Rates and Readmission Rates in Elective Colorectal Surgery. Ann Surg. 2015 Jun;261(6):1034-40. doi: 10.1097/SLA.0000000000001125. PMID 25607761
- [Background] Tremlett H, Fadrosh DW, Faruqi AA, Hart J, Roalstad S, Graves J, Lynch S, Waubant E; US Network of Pediatric MS Centers. Gut microbiota composition and relapse risk in pediatric MS: A pilot study. J Neurol Sci. 2016 Apr 15;363:153-7. doi: 10.1016/j.jns.2016.02.042. Epub 2016 Feb 20. PMID 27000242
- [Background] Ochoa-Reparaz J, Magori K, Kasper LH. The chicken or the egg dilemma: intestinal dysbiosis in multiple sclerosis. Ann Transl Med. 2017 Mar;5(6):145. doi: 10.21037/atm.2017.01.18. PMID 28462225
- [Background] Smits LP, Bouter KE, de Vos WM, Borody TJ, Nieuwdorp M. Therapeutic potential of fecal microbiota transplantation. Gastroenterology. 2013 Nov;145(5):946-53. doi: 10.1053/j.gastro.2013.08.058. Epub 2013 Sep 7. PMID 24018052
- [Background] Jangi S, Gandhi R, Cox LM, Li N, von Glehn F, Yan R, Patel B, Mazzola MA, Liu S, Glanz BL, Cook S, Tankou S, Stuart F, Melo K, Nejad P, Smith K, Topcuolu BD, Holden J, Kivisakk P, Chitnis T, De Jager PL, Quintana FJ, Gerber GK, Bry L, Weiner HL. Alterations of the human gut microbiome in multiple sclerosis. Nat Commun. 2016 Jun 28;7:12015. doi: 10.1038/ncomms12015. PMID 27352007
- [Background] Lee CH, Steiner T, Petrof EO, Smieja M, Roscoe D, Nematallah A, Weese JS, Collins S, Moayyedi P, Crowther M, Ropeleski MJ, Jayaratne P, Higgins D, Li Y, Rau NV, Kim PT. Frozen vs Fresh Fecal Microbiota Transplantation and Clinical Resolution of Diarrhea in Patients With Recurrent Clostridium difficile Infection: A Randomized Clinical Trial. JAMA. 2016 Jan 12;315(2):142-9. doi: 10.1001/jama.2015.18098. PMID 26757463
- [Background] Uygun A, Ozturk K, Demirci H, Oger C, Avci IY, Turker T, Gulsen M. Fecal microbiota transplantation is a rescue treatment modality for refractory ulcerative colitis. Medicine (Baltimore). 2017 Apr;96(16):e6479. doi: 10.1097/MD.0000000000006479. PMID 28422836
- [Background] Bajaj JS, Kassam Z, Fagan A, Gavis EA, Liu E, Cox IJ, Kheradman R, Heuman D, Wang J, Gurry T, Williams R, Sikaroodi M, Fuchs M, Alm E, John B, Thacker LR, Riva A, Smith M, Taylor-Robinson SD, Gillevet PM. Fecal microbiota transplant from a rational stool donor improves hepatic encephalopathy: A randomized clinical trial. Hepatology. 2017 Dec;66(6):1727-1738. doi: 10.1002/hep.29306. Epub 2017 Oct 30. PMID 28586116

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening period
Groups:
- Interventional FMT Treatment Arm: After providing written informed consent, subjects underwent screening and baseline assessments of stool and blood sampling, questionnaires, physical examination, MS rating scales, and MRI. Subjects then initiated an oral antibiotic regimen for 5 days to precondition the gut for the Fecal Microbiota Transplantation (FMT) of FMP30 donor stool and try to optimize engraftment of the FMP30 donor stool microbiome. Following standard bowel preparation for colonoscopy, subjects underwent the FMT procedure by an experienced gastroenterologist. Subjects returned for scheduled assessments and follow-up MRI for 12 weeks, with additional safety and biomarker follow-up for 36 weeks.
  FMP30 Donor Stool: FMP30 was manufactured by the non-profit stool bank Openbiome. Each FMP30 filtered donor stool engraftment has approximately 12.5g of stool per 30mL of normal saline. It is homogenized in sterile normal saline.
  Fecal Microbiota Transplantation (FMT) of FMP30 Donor Stool: Three doses of filtered donor stool engraftments homogenized in sterile normal saline (FMP30) obtained from the non-profit stool bank OpenBiome were administered via colonoscopy.
- Observational Control Arm: Subjects, who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures.
  After providing written informed consent, subjects will undergo screening and baseline assessments, including collection of blood and stool samples, demographic data collection, concomitant medication review, and an MS Relapse assessment. At week 2, subjects will mail in stool samples with a prepaid air bill and packaging. Weeks 4, 8, and 12 assessments will include concomitant medication review, relapse assessment, and blood and stool collection.
  The duration of the study for the observational control arm will last for 12 weeks. All study procedures will be performed at the University of California, San Francisco.
  Observational Control: Subjects, who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures.
Period: Overall Study
Arm/Group | Interventional FMT Treatment Arm | Observational Control Arm
Started | 4 | 1
Completed | 4 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 4 participants were recruited for the interventional arm and 1 for the observational control arm.
Groups:
- Interventional FMT Treatment Arm: After providing written informed consent, participants underwent screening and baseline assessments of stool and blood sampling, questionnaires, physical examination, MS rating scales, and MRI. Participants then initiated an oral antibiotic regimen for 5 days to precondition the gut for the Fecal Microbiota Transplantation (FMT) of FMP30 donor stool and try to optimize engraftment of the FMP30 donor stool microbiome. Following standard bowel preparation for colonoscopy, participants underwent the FMT procedure by an experienced gastroenterologist. Participants returned for scheduled assessments and follow-up MRI for 12 weeks, with additional safety and biomarker follow-up for 36 weeks.
  FMP30 Donor Stool: FMP30 was manufactured by the non-profit stool bank Openbiome. Each FMP30 filtered donor stool engraftment has approximately 12.5g of stool per 30mL of normal saline. It is homogenized in sterile normal saline.
  Fecal Microbiota Transplantation (FMT) of FMP30 Donor Stool: Three doses of filtered donor stool engraftments homogenized in sterile normal saline (FMP30) obtained from the non-profit stool bank OpenBiome were administered via colonoscopy.
- Observational Control Arm: Participants, who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures.
  After providing written informed consent, participants will undergo screening and baseline assessments, including collection of blood and stool samples, demographic data collection, concomitant medication review, and an MS Relapse assessment. At week 2, participants will mail in stool samples with a prepaid air bill and packaging. Weeks 4, 8, and 12 assessments will include concomitant medication review, relapse assessment, and blood and stool collection.
  The duration of the study for the observational control arm will last for 12 weeks. All study procedures will be performed at the University of California, San Francisco.
  Observational Control: Participants, who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration, and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures.
- Total: Total of all reporting groups
Arm/Group | Interventional FMT Treatment Arm | Observational Control Arm | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Continuous [Mean (Full Range); unit: years] | 41.5 [27 to 55] | 53 [53 to 53] | 43.8 [27 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Complete the Study Protocol
Description: This includes the proportion of participants who completed the study protocol, including the completion of the study visits at baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks, and a safety follow-up through week 48.
Time Frame: Baseline through week 48
Population: All enrolled participants who received FMT completed the study protocol; however, the study was interrupted due to the COVID-19 pandemic and a hold on the source material, and was subsequently closed to further enrollment.
Measure: Count of Participants; unit: Participants
Groups:
- Observational Control Arm: Participants, who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures.
  After providing written informed consent, participants will undergo screening and baseline assessments, including collection of blood and stool samples, demographic data collection, concomitant medication review, and an MS Relapse assessment. At week 2, participants will mail in stool samples with a prepaid air bill and packaging. Weeks 4, 8, and 12 assessments will include concomitant medication review, relapse assessment, and blood and stool collection.
  The duration of the study for the observational control arm will last for 12 weeks. All study procedures will be performed at the University of California, San Francisco.
  Observational Control: Participants, who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures.
Arm/Group | Interventional FMT Treatment Arm | Observational Control Arm
Number analyzed (Participants) | 4 | 1
Participants | 4 | 1

2. Primary Outcome: Change in Fecal Microbiota
Description: Engraftment: Change in fecal microbiota community structure at Baseline Visit, 2 weeks, 4 weeks, 8 weeks, 12 weeks by 16S ribosomal RNA amplicon sequencing (as a measure of the diversity of fecal microbiota by detecting sequence variations).
  Comment on unit of measure: The Shannon Index is used to assess changes in fecal microbiota diversity, with higher values indicating greater microbial diversity. Changes in the Shannon index over time will reflect the impact of the intervention on gut microbial composition.
Time Frame: Baseline Visit, 2 weeks, 4 weeks, 8 weeks, and 12 weeks.
Population: No samples were collected for the control participant at any of the time points ( Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks) as the study was interrupted due to COVID-19. We don't have data to report for the change in microbiota structure for the control participant, who did not receive an intervention. This data will also not be reported in the future (as it was not collected).
Measure: Number; unit: Shannon index
Groups:
- Change in Microbiota Structure at Baseline in FMT Treatment Arm; Change in Microbiota Structure at Week 2 in FMT Treatment Arm; Change in Microbiota Structure at Week 4 in FMT Treatment Arm; Change in Microbiota Structure at Week 8 in FMT Treatment Arm; Change in Microbiota Structure at Week 12 in FMT Treatment Arm: After providing written informed consent, participants underwent screening and baseline assessments of stool and blood sampling, questionnaires, physical examination, MS rating scales, and MRI. Participants then initiated an oral antibiotic regimen for 5 days to precondition the gut for the Fecal Microbiota Transplantation (FMT) of FMP30 donor stool and try to optimize engraftment of the FMP30 donor stool microbiome. Following standard bowel preparation for colonoscopy, participants underwent the FMT procedure by an experienced gastroenterologist. Participants returned for scheduled assessments and follow-up MRI for 12 weeks, with additional safety and biomarker follow-up for 36 weeks.
  FMP30 Donor Stool: FMP30 was manufactured by the non-profit stool bank Openbiome. Each FMP30 filtered donor stool engraftment has approximately 12.5g of stool per 30mL of normal saline. It is homogenized in sterile normal saline.
  Fecal Microbiota Transplantation (FMT) of FMP30 Donor Stool: Three doses of filtered donor stool engraftments homogenized in sterile normal saline (FMP30) obtained from the non-profit stool bank OpenBiome were administered via colonoscopy.
Arm/Group | Change in Microbiota Structure at Baseline in FMT Treatment Arm | Change in Microbiota Structure at Week 2 in FMT Treatment Arm | Change in Microbiota Structure at Week 4 in FMT Treatment Arm | Change in Microbiota Structure at Week 8 in FMT Treatment Arm | Change in Microbiota Structure at Week 12 in FMT Treatment Arm
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
Shannon index
  Participant 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Participant 1 | 0.87 | 4.60 | 4.10 | 4.50 | 4.10
  Participant 2: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Participant 2 | 1.10 | 5.78 | 5.70 | 5.80 | 5.85
  Participant 3: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Participant 3 | 5.10 | 5.60 | 5.15 | 5.18 | 5.20
  Participant 4: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Participant 4 | 2.35 | 3.90 | 3.85 | 3.95 | 3.80

3. Primary Outcome: Number of Treatment-Emergent Serious Adverse Events [Safety and Tolerability]
Description: Treatment-emergent serious adverse events from baseline through week 12. The proportion of participants who develop an adverse event (AE) of severity grade 2 or more by NIH CTCAE criteria V4.0 is considered serious. NIH CTCAE is a standardized classification and severity grading scale for adverse events used in clinical trials. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE. Grade 1 is considered mild, Grade 2 as moderate, Grade 3 as severe or medically significant, Grade 4 as life-threatening, and Grade 5 as death related to AE.
Time Frame: Baseline Visit, 2 weeks, 4 weeks, 8 weeks, and 12 weeks.
Population: All participants were monitored for the number of treatment-emergent serious adverse events from baseline through week 12.
Measure: Number; unit: number of events
Groups:
- Number of Serious AE at Baseline; Number of Serious AE at Week 2; Number of Serious AE at Week 4; Number of Serious AE at Week 8; Number of Serious AE at Week 12: Interventional arm:
  After providing written informed consent, subjects underwent screening and baseline assessments of stool and blood sampling, questionnaires, physical examination, MS rating scales, and MRI. Subjects then initiated an oral antibiotic regimen for 5 days to precondition the gut for the Fecal Microbiota Transplantation (FMT) of FMP30 donor stool and try to optimize engraftment of the FMP30 donor stool microbiome. Following standard bowel preparation for colonoscopy, subjects underwent the FMT procedure by an experienced gastroenterologist.
  FMP30 Donor Stool: FMP30 was manufactured by the non-profit stool bank Openbiome. Each FMP30 filtered donor stool engraftment has approximately 12.5g of stool per 30mL of normal saline. It is homogenized in sterile normal saline.
  Fecal Microbiota Transplantation (FMT) of FMP30 Donor Stool: Three doses of filtered donor stool engraftments homogenized in sterile normal saline (FMP30) obtained from the non-profit stool bank OpenBiome were administered via colonoscopy.
  Observational arm:
  Participants, who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures.
Arm/Group | Number of Serious AE at Baseline | Number of Serious AE at Week 2 | Number of Serious AE at Week 4 | Number of Serious AE at Week 8 | Number of Serious AE at Week 12
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
number of events
  Interventional arm: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
  Interventional arm | 0 | 0 | 0 | 0 | 0
  Observational arm: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Observational arm | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Treatment-Emergent Non-Serious Adverse Events [Safety and Tolerability]
Description: Treatment-emergent non-serious adverse events from baseline through week 12. The proportion of participants who develop an adverse event (AE) of severity grade 2 or more by NIH CTCAE criteria V4.0 is considered serious. NIH CTCAE is a standardized classification and severity grading scale for adverse events used in clinical trials. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE. Grade 1 is considered mild, Grade 2 as moderate, Grade 3 as severe or medically significant, Grade 4 as life-threatening, and Grade 5 as death related to AE.
Time Frame: Baseline Visit, 2 weeks, 4 weeks, 8 weeks, and 12 weeks.
Population: All participants were monitored for the number of treatment-emergent non-serious adverse events from baseline through week 12.
Measure: Number; unit: Number of events
Groups:
- Number of Non-serious AE at Baseline; Number of Non-serious AE at Week 2; Number of Non-serious AE at Week 4; Number of Non-serious AE at Week 8; Number of Non-serious AE at Week 12: Interventional arm:
  After providing written informed consent, subjects underwent screening and baseline assessments of stool and blood sampling, questionnaires, physical examination, MS rating scales, and MRI. Subjects then initiated an oral antibiotic regimen for 5 days to precondition the gut for the Fecal Microbiota Transplantation (FMT) of FMP30 donor stool and try to optimize engraftment of the FMP30 donor stool microbiome. Following standard bowel preparation for colonoscopy, subjects underwent the FMT procedure by an experienced gastroenterologist.
  FMP30 Donor Stool: FMP30 was manufactured by the non-profit stool bank Openbiome. Each FMP30 filtered donor stool engraftment has approximately 12.5g of stool per 30mL of normal saline. It is homogenized in sterile normal saline.
  Fecal Microbiota Transplantation (FMT) of FMP30 Donor Stool: Three doses of filtered donor stool engraftments homogenized in sterile normal saline (FMP30) obtained from the non-profit stool bank OpenBiome were administered via colonoscopy.
  Observational arm:
  Participants, who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration, and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures.
Arm/Group | Number of Non-serious AE at Baseline | Number of Non-serious AE at Week 2 | Number of Non-serious AE at Week 4 | Number of Non-serious AE at Week 8 | Number of Non-serious AE at Week 12
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
Number of events
  Interventional arm: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
  Interventional arm | 1 | 0 | 0 | 0 | 0
  Observational arm: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Observational arm | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Change in Plasma CD19+ B Cells in Interventional Arm [CD19: Cluster of Differentiation Antigen 19]
Description: Plasma CD19+ B cell count will be measured as absolute cell counts (cells/uL) at Baseline Visit, 2 weeks, 4 weeks, 8 weeks, and 12 weeks.
Time Frame: Baseline Visit, 2 weeks, 4 weeks, 8 weeks, and 12 weeks.
Population: Plasma CD19+ cell counts were measured at Weeks 0, 2, 4, 8, and 12. Some participants were not able to complete the visit due to the COVID-19 pandemic; therefore, the number of participants analyzed is 0.
Measure: Number; unit: cells/uL
Groups:
- Absolute B-cell Count at Baseline; Absolute B-cell Count at Week 2; Absolute B-cell Count at Week 4; Absolute B-cell Count at Week 8; Absolute B-cell Count at Week 12: Interventional arm:
  After providing written informed consent, subjects underwent screening and baseline assessments of stool and blood sampling, questionnaires, physical examination, MS rating scales, and MRI. Subjects then initiated an oral antibiotic regimen for 5 days to precondition the gut for the Fecal Microbiota Transplantation (FMT) of FMP30 donor stool and try to optimize engraftment of the FMP30 donor stool microbiome. Following standard bowel preparation for colonoscopy, subjects underwent the FMT procedure by an experienced gastroenterologist.
  FMP30 Donor Stool: FMP30 was manufactured by the non-profit stool bank Openbiome. Each FMP30 filtered donor stool engraftment has approximately 12.5g of stool per 30mL of normal saline. It is homogenized in sterile normal saline.
  Fecal Microbiota Transplantation (FMT) of FMP30 Donor Stool: Three doses of filtered donor stool engraftments homogenized in sterile normal saline (FMP30) obtained from the non-profit stool bank OpenBiome were administered via colonoscopy.
Arm/Group | Absolute B-cell Count at Baseline | Absolute B-cell Count at Week 2 | Absolute B-cell Count at Week 4 | Absolute B-cell Count at Week 8 | Absolute B-cell Count at Week 12
Number analyzed (Participants) | 4 | 4 | 2 | 4 | 3
cells/uL
  Participant 1: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1
  Participant 1 | 210 | 276 |  | 204 | 245
  Participant 2: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Participant 2 | 133 | 139 | 137 | 143 | 130
  Participant 3: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Participant 3 | 269 | 218 | 168 | 220 | 217
  Participant 4: number analyzed (Participants) | 1 | 1 | 0 | 1 | 0
  Participant 4 | 55 | 65 |  | 74 |

6. Secondary Outcome: Change in Plasma CD19+ B Cells in Observational Arm
Description: as for outcome 5
Time Frame: Baseline Visit, 2 weeks, 4 weeks, 8 weeks, and 12 weeks.
Population: as for outcome 5
Measure: Number; unit: cells/uL
Groups:
- Absolute B-cell Count at Baseline; Absolute B-cell Count at Week 2; Absolute B-cell Count at Week 4; Absolute B-cell Count at Week 8; Absolute B-cell Count at Week 12: Observational Arm:
  Participants, who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration, and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures
Arm/Group | Absolute B-cell Count at Baseline | Absolute B-cell Count at Week 2 | Absolute B-cell Count at Week 4 | Absolute B-cell Count at Week 8 | Absolute B-cell Count at Week 12
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 1
cells/uL | 198 |  | 195 | 214 | 178

7. Secondary Outcome: Change in Serum IgA Immunoglobulin Levels in Interventional Arm [IgA: Immunoglobulin A]
Description: Serum Immunoglobulin levels of IgA will be measured in mg/dL at Baseline Visit, 2 weeks, 4 weeks, 8 weeks, and 12 weeks.
Time Frame: Baseline Visit, 2 weeks, 4 weeks, 8 weeks, and 12 weeks.
Population: Serum immunoglobulin levels at Weeks 0, 2, 4, 8, and 12 were collected. Some participants were not able to complete the visit due to the COVID-19 pandemic; therefore, the number of participants analyzed is 0.
Measure: Number; unit: mg/dL
Groups:
- Serum IgA Level at Baseline; Serum IgA Level at 2 Weeks; Serum IgA Level at 4 Weeks; Serum IgA Level at 8 Weeks; Serum IgA Level at 12 Weeks: Interventional arm:
  After providing written informed consent, subjects underwent screening and baseline assessments of stool and blood sampling, questionnaires, physical examination, MS rating scales, and MRI. Subjects then initiated an oral antibiotic regimen for 5 days to precondition the gut for the Fecal Microbiota Transplantation (FMT) of FMP30 donor stool and try to optimize engraftment of the FMP30 donor stool microbiome. Following standard bowel preparation for colonoscopy, subjects underwent the FMT procedure by an experienced gastroenterologist.
  FMP30 Donor Stool: FMP30 was manufactured by the non-profit stool bank Openbiome. Each FMP30 filtered donor stool engraftment has approximately 12.5g of stool per 30mL of normal saline. It is homogenized in sterile normal saline.
  Fecal Microbiota Transplantation (FMT) of FMP30 Donor Stool: Three doses of filtered donor stool engraftments homogenized in sterile normal saline (FMP30) obtained from the non-profit stool bank OpenBiome were administered via colonoscopy.
Arm/Group | Serum IgA Level at Baseline | Serum IgA Level at 2 Weeks | Serum IgA Level at 4 Weeks | Serum IgA Level at 8 Weeks | Serum IgA Level at 12 Weeks
Number analyzed (Participants) | 4 | 4 | 2 | 4 | 4
mg/dL
  Participant 1: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1
  Participant 1 | 89 | 90 |  | 79 | 137
  Participant 2: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Participant 2 | 129 | 117 | 127 | 120 | 128
  Participant 3: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Participant 3 | 381 | 387 | 397 | 337 | 380
  Participant 4: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1
  Participant 4 | 248 | 221 |  | 253 | 236

8. Secondary Outcome: Change in Serum IgA Immunoglobulin Levels in Observational Arm
Description: Serum Immunoglobulin levels of IgA will be measured in mg/dL at Baseline Visit, 2 weeks, 4 weeks, and 12 weeks.
Time Frame: Baseline Visit, 2 weeks, 4 weeks, and 12 weeks.
Population: as for outcome 7
Measure: Number; unit: mg/dL
Groups:
- Serum IgA Level at Baseline; Serum IgA Level at 2 Weeks; Serum IgA Level at 4 Weeks; Serum IgA Level at 8 Weeks; Serum IgA Level at 12 Weeks: Observational Arm:
  Participants, who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures.
Arm/Group | Serum IgA Level at Baseline | Serum IgA Level at 2 Weeks | Serum IgA Level at 4 Weeks | Serum IgA Level at 8 Weeks | Serum IgA Level at 12 Weeks
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 1
mg/dL |  |  | 647 | 589 | 579

9. Secondary Outcome: Change in Serum IgM Immunoglobulin Levels in Interventional Arm [IgM: Immunoglobulin M]
Description: Serum Immunoglobulin levels of IgM will be measured in mg/dL at Baseline Visit, 2 weeks, 4 weeks, 8 weeks, and 12 weeks.
Time Frame: Baseline Visit, 2 weeks, 4 weeks, 8 weeks and 12 weeks.
Population: as for outcome 7
Measure: Number; unit: mg/dL
Groups:
- Serum IgM Level at Baseline; Serum IgM Level at 2 Weeks; Serum IgM Level at 4 Weeks; Serum IgM Level at 8 Weeks; Serum IgM Level at 12 Weeks: Interventional arm:
  After providing written informed consent, subjects underwent screening and baseline assessments of stool and blood sampling, questionnaires, physical examination, MS rating scales, and MRI. Subjects then initiated an oral antibiotic regimen for 5 days to precondition the gut for the Fecal Microbiota Transplantation (FMT) of FMP30 donor stool and try to optimize engraftment of the FMP30 donor stool microbiome. Following standard bowel preparation for colonoscopy, subjects underwent the FMT procedure by an experienced gastroenterologist.
  FMP30 Donor Stool: FMP30 was manufactured by the non-profit stool bank Openbiome. Each FMP30 filtered donor stool engraftment has approximately 12.5g of stool per 30mL of normal saline. It is homogenized in sterile normal saline.
  Fecal Microbiota Transplantation (FMT) of FMP30 Donor Stool: Three doses of filtered donor stool engraftments homogenized in sterile normal saline (FMP30) obtained from the non-profit stool bank OpenBiome were administered via colonoscopy.
Arm/Group | Serum IgM Level at Baseline | Serum IgM Level at 2 Weeks | Serum IgM Level at 4 Weeks | Serum IgM Level at 8 Weeks | Serum IgM Level at 12 Weeks
Number analyzed (Participants) | 4 | 4 | 2 | 4 | 4
mg/dL
  Participant 1: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1
  Participant 1 | 110 | 111 |  | 99 | 112
  Participant 2: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Participant 2 | 110 | 103 | 114 | 118 | 115
  Participant 3: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Participant 3 | 77 | 79 | 82 | 69 | 81
  Participant 4: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1
  Participant 4 | 285 | 260 |  | 290 | 274

10. Secondary Outcome: Change in Serum IgM Immunoglobulin Levels in Observational Arm
Description: Serum Immunoglobulin levels of IgM will be measured in mg/dL at Baseline Visit, 2 weeks, 4 weeks, 8 weeks, and 12 weeks. The percentage of change from baseline for each time point is also reported.
Time Frame: Baseline Visit, 2 weeks, 4 weeks, 8 weeks and 12 weeks.
Population: as for outcome 7
Measure: Number; unit: mg/dL
Groups:
- Serum IgM Level at Baseline; Serum IgM Level at 2 Weeks; Serum IgM Level at 4 Weeks; Serum IgM Level at 8 Weeks; Serum IgM Level at 12 Weeks: Observational Arm:
  Participants, who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures.
Arm/Group | Serum IgM Level at Baseline | Serum IgM Level at 2 Weeks | Serum IgM Level at 4 Weeks | Serum IgM Level at 8 Weeks | Serum IgM Level at 12 Weeks
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
mg/dL |  |  | 135 |  |

11. Secondary Outcome: Change in Serum IgG Immunoglobulin Levels in Interventional Arm [IgG: Immunoglobulin G]
Description: Serum Immunoglobulin levels of IgG will be measured in mg/dL at Baseline Visit, 2 weeks, 4 weeks, 8 weeks, and 12 weeks.
Time Frame: Baseline Visit, 2 weeks, 4 weeks, 8 weeks and 12 weeks
Population: as for outcome 7
Measure: Number; unit: mg/dL
Groups:
- Serum IgG Level at Baseline; Serum IgG Level at 2 Weeks; Serum IgG Level at 4 Weeks; Serum IgG Level at 8 Weeks; Serum IgG Level at 12 Weeks: Interventional arm:
  After providing written informed consent, subjects underwent screening and baseline assessments of stool and blood sampling, questionnaires, physical examination, MS rating scales, and MRI. Subjects then initiated an oral antibiotic regimen for 5 days to precondition the gut for the Fecal Microbiota Transplantation (FMT) of FMP30 donor stool and try to optimize engraftment of the FMP30 donor stool microbiome. Following standard bowel preparation for colonoscopy, subjects underwent the FMT procedure by an experienced gastroenterologist.
  FMP30 Donor Stool: FMP30 was manufactured by the non-profit stool bank Openbiome. Each FMP30 filtered donor stool engraftment has approximately 12.5g of stool per 30mL of normal saline. It is homogenized in sterile normal saline.
  Fecal Microbiota Transplantation (FMT) of FMP30 Donor Stool: Three doses of filtered donor stool engraftments homogenized in sterile normal saline (FMP30) obtained from the non-profit stool bank OpenBiome were administered via colonoscopy.
Arm/Group | Serum IgG Level at Baseline | Serum IgG Level at 2 Weeks | Serum IgG Level at 4 Weeks | Serum IgG Level at 8 Weeks | Serum IgG Level at 12 Weeks
Number analyzed (Participants) | 4 | 4 | 2 | 4 | 4
mg/dL
  Participant 1: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1
  Participant 1 | 966 | 979 |  | 925 | 1630
  Participant 2: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Participant 2 | 1070 | 1020 | 966 | 1040 | 1100
  Participant 3: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Participant 3 | 1170 | 1250 | 1290 | 1130 | 1160
  Participant 4: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1
  Participant 4 | 939 | 855 |  | 972 | 960

12. Secondary Outcome: Change in Serum IgG Immunoglobulin Levels in Observational Arm
Description: Serum Immunoglobulin levels of IgG will be measured in mg/dL at Baseline Visit, 2 weeks, 4 weeks, 8 weeks, and 12 weeks.
Time Frame: Baseline Visit, 2 weeks, 4 weeks, 8 weeks and 12 weeks
Population: as for outcome 7
Measure: Number; unit: mg/dL
Groups:
- Serum IgG Level at Baseline; Serum IgG Level at 2 Weeks; Serum IgG Level at 4 Weeks; Serum IgG Level at 8 Weeks; Serum IgG Level at 12 Weeks: Observational Arm:
  Participants, who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures.
Arm/Group | Serum IgG Level at Baseline | Serum IgG Level at 2 Weeks | Serum IgG Level at 4 Weeks | Serum IgG Level at 8 Weeks | Serum IgG Level at 12 Weeks
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 1
mg/dL |  |  | 984 | 928 | 870

13. Secondary Outcome: Incidence of New T2/FLAIR Lesions
Description: The number of new or enlarging T2/FLAIR lesions will be counted at pre-treatment and week 12.
Time Frame: At pre-treatment visit and week 12.
Population: After screening, participants undergo MRI at pre-treatment and at Week 12 to assess for any new T2/FLAIR lesions during the treatment period in both the interventional and observational arms.
Measure: Number; unit: number of lesions
Groups:
- Number of New T2/FLAIR Lesions at Pre-treatment; Number of New T2/FLAIR Lesions at Week 12: Interventional arm:
  After providing written informed consent, subjects underwent screening and baseline assessments of stool and blood sampling, questionnaires, physical examination, MS rating scales, and MRI. Subjects then initiated an oral antibiotic regimen for 5 days to precondition the gut for the Fecal Microbiota Transplantation (FMT) of FMP30 donor stool and try to optimize engraftment of the FMP30 donor stool microbiome. Following standard bowel preparation for colonoscopy, subjects underwent the FMT procedure by an experienced gastroenterologist.
  FMP30 Donor Stool: FMP30 was manufactured by the non-profit stool bank Openbiome. Each FMP30 filtered donor stool engraftment has approximately 12.5g of stool per 30mL of normal saline. It is homogenized in sterile normal saline.
  Fecal Microbiota Transplantation (FMT) of FMP30 Donor Stool: Three doses of filtered donor stool engraftments homogenized in sterile normal saline (FMP30) obtained from the non-profit stool bank OpenBiome were administered via colonoscopy.
  Observational arm:
  Participants, who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration, and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures.
Arm/Group | Number of New T2/FLAIR Lesions at Pre-treatment | Number of New T2/FLAIR Lesions at Week 12
Number analyzed (Participants) | 5 | 5
number of lesions
  Interventional arm: number analyzed (Participants) | 4 | 4
  Interventional arm | 0 | 1
  Observational arm: number analyzed (Participants) | 1 | 1
  Observational arm | 0 | 0

14. Secondary Outcome: Treatment-emergent Gadolinium Enhancing Lesions
Description: New treatment-emergent gadolinium-enhancing lesions on brain MRI.
Time Frame: At pre-treatment visit and week 12.
Population: After screening, participants undergo MRI at pre-treatment and at Week 12 to assess for any new enhancing lesions in both the interventional and observational arms.
Measure: Number; unit: number of enhancing lesions
Groups:
- Treatment-emergent Gadolinium-Enhancing Lesions at Pre-treatment; Treatment-emergent Gadolinium-Enhancing Lesions at Week 12: Interventional arm:
  After providing written informed consent, subjects underwent screening and baseline assessments of stool and blood sampling, questionnaires, physical examination, MS rating scales, and MRI. Subjects then initiated an oral antibiotic regimen for 5 days to precondition the gut for the Fecal Microbiota Transplantation (FMT) of FMP30 donor stool and try to optimize engraftment of the FMP30 donor stool microbiome. Following standard bowel preparation for colonoscopy, subjects underwent the FMT procedure by an experienced gastroenterologist.
  FMP30 Donor Stool: FMP30 was manufactured by the non-profit stool bank Openbiome. Each FMP30 filtered donor stool engraftment has approximately 12.5g of stool per 30mL of normal saline. It is homogenized in sterile normal saline.
  Fecal Microbiota Transplantation (FMT) of FMP30 Donor Stool: Three doses of filtered donor stool engraftments homogenized in sterile normal saline (FMP30) obtained from the non-profit stool bank OpenBiome were administered via colonoscopy.
  Observational arm:
  Participants, who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration, and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures.
Arm/Group | Treatment-emergent Gadolinium-Enhancing Lesions at Pre-treatment | Treatment-emergent Gadolinium-Enhancing Lesions at Week 12
Number analyzed (Participants) | 5 | 5
number of enhancing lesions
  Interventional arm: number analyzed (Participants) | 4 | 4
  Interventional arm | 0 | 1
  Observational arm: number analyzed (Participants) | 1 | 1
  Observational arm | 0 | 0

15. Secondary Outcome: Clinical Relapse
Description: Clinical relapse through week 12 (treatment phase)
Time Frame: From baseline to week 12
Population: Participants were monitored for clinical relapse through week 12.
Measure: Number; unit: Number of clinical relapses
Groups:
- Observational Control Arm: Subjects, who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures.
  After providing written informed consent, subjects will undergo screening and baseline assessments, including collection of blood and stool samples, demographic data collection, concomitant medication review, and an MS Relapse assessment. At week 2, subjects will mail in stool samples with a prepaid air bill and packaging. Weeks 4, 8, and 12 assessments will include concomitant medication review, relapse assessment, and blood and stool collection.
  The duration of the study for the observational control arm will last for 12 weeks. All study procedures will be performed at the University of California, San Francisco.
  Participants were monitored for clinical relapse through week 12.
Arm/Group | Interventional FMT Treatment Arm | Observational Control Arm
Number analyzed (Participants) | 4 | 1
Number of clinical relapses | 0 | 0

16. Secondary Outcome: Percentage of Induced T-regulatory Cells
Description: Flow cytometric analysis of peripheral blood mononuclear cells (PBMC) from each participant and at each time point. T-regs were induced by stimulation of PBMCs with anti-CD3 and anti-CD28 antibodies in the presence of IL2 and TGFb. The percentage of T-regs before and after FMT was analyzed. FMT was performed during the baseline visit. [CD3: cluster of differentiation 3, CD28: cluster of differentiation 28, IL2: interleukin2, TGFb: Transforming growth factor beta]
Time Frame: Pre-screening, Screening, Baseline, Week 2, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48
Population: Participants who completed the treatment arm were assessed for changes in fecal microbiota using 16S ribosomal RNA sequencing. Per the study protocol, no FMT intervention was performed in participants from the observation arm; therefore, only participants in the interventional arm are included in this secondary outcome analysis. Some participants were not able to complete the visit due to the COVID-19 pandemic; therefore, the number of participants analyzed is 0.
Measure: Number; unit: percentage of T-regs
Groups:
- Average Percentage of Induced T-regs at Pre-screening; Average Percentage of Induced T-regs at Screening; Average Percentage of Induced T-regs at Baseline; Average Percentage of Induced T-regs at 2 Weeks; Average Percentage of Induced T-regs Level at 4 Weeks; Average Percentage of Induced T-regs at 8 Weeks; Average Percentage of Induced T-regs at 12 Weeks; Average Percentage of Induced T-regs at 24 Weeks; Average Percentage of Induced T-regs at 36 Weeks; Average Percentage of Induced T-regs at Week 48: Interventional arm:
  After providing written informed consent, subjects underwent screening and baseline assessments of stool and blood sampling, questionnaires, physical examination, MS rating scales, and MRI. Subjects then initiated an oral antibiotic regimen for 5 days to precondition the gut for the Fecal Microbiota Transplantation (FMT) of FMP30 donor stool and try to optimize engraftment of the FMP30 donor stool microbiome. Following standard bowel preparation for colonoscopy, subjects underwent the FMT procedure by an experienced gastroenterologist. Subjects returned for scheduled assessments and follow-up MRI for 12 weeks, with additional safety and biomarker follow-up for 36 weeks.
  FMP30 Donor Stool: FMP30 was manufactured by the non-profit stool bank Openbiome. Each FMP30 filtered donor stool engraftment has approximately 12.5g of stool per 30mL of normal saline. It is homogenized in sterile normal saline.
Arm/Group | Average Percentage of Induced T-regs at Pre-screening | Average Percentage of Induced T-regs at Screening | Average Percentage of Induced T-regs at Baseline | Average Percentage of Induced T-regs at 2 Weeks | Average Percentage of Induced T-regs Level at 4 Weeks | Average Percentage of Induced T-regs at 8 Weeks | Average Percentage of Induced T-regs at 12 Weeks | Average Percentage of Induced T-regs at 24 Weeks | Average Percentage of Induced T-regs at 36 Weeks | Average Percentage of Induced T-regs at Week 48
Number analyzed (Participants) | 4 | 2 | 4 | 2 | 4 | 3 | 4 | 3 | 3 | 3
percentage of T-regs
  Participant 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
  Participant 1 | 24.8 | 21.1 | 18.4 | 23.8 | 22.9 | 17.2 | 14.8 | 20.7 | 20.8 | 13.2
  Participant 2: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
  Participant 2 | 23.5 | 25.1 | 20.1 | 25.3 | 25.6 | 21.4 | 19.8 | 18.2 | 18.0 | 16.6
  Participant 3: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1
  Participant 3 | 15.2 |  | 24.5 |  | 24.7 | 22.4 | 19.7 | 19.7 | 17.0 | 15.6
  Participant 4: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Participant 4 | 21.5 |  | 14.5 |  | 12.2 |  | 12.4 |  |  |

ADVERSE EVENTS:
Time Frame: 12-week treatment phase (FMT) and 36-week safety follow-up for the interventional arm, and 12 weeks for the observational arm.
Description: The proportion of participants who develop an adverse event (AE) of severity grade 2 or more by NIH CTCAE criteria V4.0 is considered serious. NIH CTCAE is a standardized classification and severity grading scale used for AEs in clinical trials. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE. Grade 1 is considered mild, Grade 2 as moderate, Grade 3 as severe or medically significant, Grade 4 as life-threatening, and Grade 5 as death related to AE.
Groups:
- Number of Events at 12 Weeks for Interventional FMT Treatment Arm; Number of Events at 36 Weeks for Interventional FMT Treatment Arm: After providing written informed consent, participants underwent screening and baseline assessments of stool and blood sampling, questionnaires, physical examination, MS rating scales, and MRI. Participants then initiated an oral antibiotic regimen for 5 days to precondition the gut for the Fecal Microbiota Transplantation (FMT) of FMP30 donor stool and try to optimize engraftment of the FMP30 donor stool microbiome. Following standard bowel preparation for colonoscopy, participants underwent the FMT procedure by an experienced gastroenterologist. Participants returned for scheduled assessments and follow-up MRI for 12 weeks, with additional safety and biomarker follow-up for 36 weeks.
  FMP30 Donor Stool: FMP30 was manufactured by the non-profit stool bank Openbiome. Each FMP30 filtered donor stool engraftment has approximately 12.5g of stool per 30mL of normal saline. It is homogenized in sterile normal saline.
  Fecal Microbiota Transplantation (FMT) of FMP30 Donor Stool: Three doses of filtered donor stool engraftments homogenized in sterile normal saline (FMP30) obtained from the non-profit stool bank OpenBiome were administered via colonoscopy.
- Number of Events at 12 Weeks for Observational Control Arm: Participants, who otherwise satisfy study inclusion criteria based on their MS phenotype, demographics, disease duration, and prior use of allowable MS therapies, will be recruited as a comparison observational group to measure stability of stool and serum immunological measures.
  After providing written informed consent, participants will undergo screening and baseline assessments, including collection of blood and stool samples, demographic data collection, concomitant medication review, and an MS Relapse assessment. At week 2, participants will mail in stool samples with a prepaid air bill and packaging. Weeks 4, 8, and 12 assessments will include concomitant medication review, relapse assessment, and blood and stool collection.
  The duration of the study for the observational control arm will last for 12 weeks. All study procedures will be performed at the University of California, San Francisco.
Arm/Group | Number of Events at 12 Weeks for Interventional FMT Treatment Arm | Number of Events at 36 Weeks for Interventional FMT Treatment Arm | Number of Events at 12 Weeks for Observational Control Arm
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Number of Events at 12 Weeks for Interventional FMT Treatment Arm (N=4) | Number of Events at 36 Weeks for Interventional FMT Treatment Arm (N=4) | Number of Events at 12 Weeks for Observational Control Arm (N=1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal cramping / stomach upset (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) — Mild, transient
Diarrhea/Loose Stool (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Dysgeusia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Drowsiness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection reaction to MS medication (General disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (General disorders) | 0 (0) | 1 (1) | 0 (0) — Grade 1, transient
Temperature regulation (felt warmer or colder) (General disorders) | 1 (1) | 0 (0) | 0 (0)
Intertrigo (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Otitis Media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spider bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
AST elevation (<2.5x normal) (Investigations) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Investigations) | 1 (1) | 0 (0) | 0 (0) — Mild, transient
Lumbar Strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Heat related worsening of neurologic symptoms (typical of MS) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Numbness / Tingling (transient) (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Scalp itch (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was not fully recruited. Study recruitment was interrupted by both the COVID-19 pandemic and a hold on the FMT source material. Participants recruited up until that point were analyzed with available safety and outcome data reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT03594487/Prot_SAP_000.pdf